CLINICAL TRIAL: NCT05194956
Title: Orthodontic Patient Experience of Intraoral Scanners Versus Alginate Impressions in the UK: a Single-Centre Randomised Controlled Crossover Trial
Brief Title: Orthodontic Patient Experience of Intraoral Scans Versus Alginate Impressions
Acronym: OPESI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Collaborators: British Orthodontic Society Foundation (Unknown); Derby Pump Priming Charitable Funds (Unknown); Derby Clinical Trials Support Unit (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UHDB/2021/022
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-12

CONDITIONS: Orthodontic Patient Experience
Keywords: Orthodontic Patient; Intraoral Scan; Alginate impression; Conventional impression; Digital scan; Patient experience; Patient comfort; Preference

STUDY DESIGN:
Intervention Model Description: Single-centre prospective randomised controlled two-period crossover study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 - Alginate impressions followed by digital intraoral scan (Experimental): The participant will have alginate impressions taken for orthodontic treatment records first. Followed by a digital intraoral scan a minimum of 4-6 weeks washout period. After each intervention, the participant will complete a modified visual analogue scale (VAS) questionnaire about their experience.
  Interventions: Procedure: Intraoral scan; Procedure: Alginate impressions
- Arm 2 - Digital intraoral scan followed by alginate impressions (Experimental): The participant will have a digital intraoral taken for orthodontic treatment records first. Followed by alginate impressions a minimum of 4-6 weeks washout period. After each intervention, the participant will complete a modified visual analogue scale (VAS) questionnaire about their experience.
  Interventions: Procedure: Intraoral scan; Procedure: Alginate impressions

INTERVENTIONS:
Procedure: Intraoral scan — An intraoral scan is multiple images taken using an intraoral scanning device which results in a digital mould being taken of the participants mouth and bite. It works by systematically placing the scanner tip over the teeth and gums, whilst it constructs an image on screen.
Procedure: Alginate impressions — Alginate impressions are the conventional method of creating dental moulds for orthodontic records. A plastic tray is filled with an alginate material, which is placed into the mouth to take a mould of the teeth. This requires two moulds for both top and bottom arches. In addition, the participant would also bite into a warm piece of wax to record their bite.

SUMMARY:
CONTEXT: Digital scanning systems are becoming more and more popular with the advent of the COVID-19 pandemic. The risks surrounding aerosol-generating procedures (AGP) has resulted in practitioners changing their normal practice and finding alternative methods to continue managing their patients. Digital (intraoral) scanners are often used to show patients treatment options and help in educating them regarding their oral hygiene as it produces an almost instant digital image of their teeth. Conventional methods using alginate impressions produce study models which are created in dental plaster or stone, involving a lab cost and a greater environmental impact but remain a popular method of recording a patient's teeth and bite.

OBJECTIVE: To investigate patient experience, operator experience and preference in intraoral scanning versus alginate impression taking in the orthodontic setting.

DESIGN, SETTING AND SUBJECTS: A randomised controlled two-period crossover trial to be conducted in a UK secondary care setting involving 84 participants ready to start orthodontic treatment, with no experience of impressions/intraoral scans in the last 2 years. Patients with cleft lip and/or palate or recent research involvement will be excluded.

OUTCOMES: A modified visual analogue scale, will be used to measure patient and operator reported outcomes (e.g. patient comfort, operator confidence, perceived time taken and induction of cough/gag reflex) following an alginate impression or an intraoral scan using Trios® 3 intraoral scanner (3Shape). The time taken for each procedure will also be measured. Lastly, operator preference will be recorded.

CONCLUSION: The proposed study aims to add to the limited evidence base, providing information regarding the use of intraoral scanners compared to alginate impressions from both the orthodontic patient and operator perspectives.

DETAILED DESCRIPTION:
Eligible patients are to be identified during a virtual dental health education (DHE) appointment prior to their orthodontic treatment commencing. With consent, the trial will be discussed with patients meeting the inclusion criteria and they will be provided with relevant trial information in both leaflet and video format. The potential participant and/or their parent or guardian will be allowed time (3 weeks) to consider the information and ask any relevant questions. If they choose to take part in the trial, they will be recruited and allocated randomly into mixed block sizes using an online randomisation tool. If they choose not to participate, normal orthodontic care will continue. For children, unable to consent for themselves, assent will also be sought.

Once the participant has provided appropriate consent/assent, the following procedure will be followed:

• One unit will be set up with an operator and a nurse

Participants in the alginate impression group:

1. The unit the participant will be treated in, will be set up appropriately with relevant materials ready.

   * The alginate to be used will be: Zhermack orthoprint® orthodontic alginate material
2. A timer will be started when the participant is seated in the chair
3. The operator will carry out the impression as normal:

   * Tray selection
   * Alginate mixing
   * Tray seating
   * Alginate setting
   * Tray removal
   * Wax bite
   * Clean up of the participant's face
4. The timer will be stopped
5. Questionnaires

   * Participant will be asked to complete a questionnaire (modified VAS using pictorial anchors)
   * Operator will be asked to complete a questionnaire
6. These will be collected for analysis
7. The participant will then have records taken as part of their normal orthodontic care, if not done already +/- a discussion to consent patient for orthodontic treatment
8. The participants will return a minimum 4 weeks later for a second appointment (if they have not had an intraoral scan already) in which they will undertake the process for 'Participants in the intraoral scanner group'

Participants in the intraoral scanner group:

1. The unit the participant will be treated in, will be set up appropriately with relevant materials ready. The interchangeable covering will be placed over the scanner ready for use.

   * The intraoral scanning device to be used will be: Trios® 3 intraoral scanner (3Shape)
   * The staff will be appropriately trained and will be requested to carry out a minimum of 10 scans prior to the study beginning
2. A timer will be started when the participant is seated in the chair
3. The scan will be carried out as per the manufacturer's directions to include a full mouth scan and bite registration and saved on the scanner system.
4. The timer will be stopped
5. Questionnaires

   * Participant will be asked to complete a questionnaire (modified VAS using pictorial anchors)
   * Operator will be asked to complete a questionnaire
6. These will be collected for analysis
7. The participant will then have records taken as part of their normal orthodontic care, if not done already +/- a discussion to consent patient for orthodontic treatment +/- fit of any orthodontic appliance required.
8. The participants will return a minimum 4 weeks later for a second appointment (if they have not had an alginate impression already) in which they will undertake the process for 'Participants in the alginate impression group'

A minimum of 4 weeks between the two appointments allows for an adequate washout period and it also fits with orthodontic laboratory work timelines within the hospital.

Once all participant data is obtained, the operators will be asked a single question to indicate their preference towards a single method.

Any participant and/or their parent or guardian, if appropriate who wishes to withdraw at any point during the trial can do so without reason and without this affecting or prejudicing the delivery of their orthodontic care.

Analyses:

* Primary outcome - the difference between the paired visual analogue scale (VAS) scores will be compared using analysis of variance (ANOVA) that will analyse the period, treatment and sequence effects of the comfort scores.
* Secondary outcomes - the 8 secondary outcomes measured by VAS and the time taken to make the impression or complete the scan will be compared using analyses of variance suitable for a crossover study, that will test the period, treatment and sequence effects on these nine secondary outcomes. The operator's preference will be reported using descriptive statistics. The frequency and percentages will be recorded.

Only the primary analysis will be compared against a specific level of significance. The secondary analyses should be considered as hypothesis generating rather than providing firm conclusions.

ELIGIBILITY:
Inclusion Criteria:

* New patients, aged 10 years and old, attending the Royal Derby Hospital orthodontic department, requiring study model impressions taken prior to commencing orthodontic treatment
* Participants must be capable of giving informed consent, or have an acceptable individual capable of giving consent on the patient's behalf (e.g. parent or guardian of a child under 16 years of age).

Exclusion Criteria:

* Patients who have had previous experience of impressions/intraoral scans in the last 2 years
* Cleft lip and/or palate patients
* Patient who have been involved in a study in the last 6 months or are currently part of a study

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Murray, BDS, MSc, FDS RCPS, MOrth RCS, Principal Investigator — University Hospitals of Derby and Burton NHS Trust
Locations (1):
- Royal Derby Hospital, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Only anonymised participant data will be shared on request e.g. for inclusion in a systematic review and meta-analysis.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study data is anticipated to become available following publication. Study data will be archived for 5 years from the end of the study.
Access Criteria: Analyses within a meta-analysis would be considered if it has been approved through an independent review committee. Requests may be submitted up to 5 years from the end of the study.

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan | Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions
Started | 42 | 44
Completed | 42 | 44
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan | Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions
Started | 42 | 44
Completed | 42 | 42
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Period 2
Arm/Group | Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan | Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions
Started | 42 | 42
Completed | 42 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The primary analysis was intended to be completed on all patients, after imputing any missing data. However, the primary analysis was carried out on complete records only, although there were 2 patients who withdrew after their first procedure. The missing data for these two patients was not imputed because the imputation of two values using multiple imputation would not add any value to the statistical analysis or results. In addition, the required sample of 84 patients had been achieved.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan | Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (4.23) | 14.1 (3.10) | 14.2 (3.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 21 | 19 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 30 | 32 | 62
  Ethnicity: Pakistani | 4 | 3 | 7
  Ethnicity: Mixed heritage | 3 | 3 | 6
  Ethnicity: Indian | 2 | 1 | 3
  Ethnicity: Black African | 0 | 1 | 1
  Ethnicity: Black Caribbean | 1 | 0 | 1
  Ethnicity: Not given | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United Kingdom | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Orthodontic Patient Comfort
Description: A 100mm modified Visual Analogue Scale (VA scale) measuring patient comfort during intraoral scanning taking versus alginate impressions taken in the orthodontic setting. A higher score would indicate a more negative experience. Minimum value: 0, Maximum value: 100
Time Frame: Immediately following intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan | Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions
Number analyzed (Participants) | 42 | 42
score on a scale | 9.2 [2.46 to 15.97] | 7.7 [0.87 to 14.51]
Statistical Analysis 1: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; All units of measure reported for this analysis are the mean within-patient differences between alginate and scan VAS scores (i.e. alginate score - scan score); Test type: Superiority; p = 0.0006, Two-period two-treatment crossover ANOVA; P-values are calculated taking sequence and period effects into account; Mean Difference (Net) = 8.5, 95% CI 2-sided [3.75 to 13.15] — This estimation value assumes period and sequence effects are equal between the treatments
Statistical Analysis 2: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Sequence effects; p = 0.1984, ANOVA
Statistical Analysis 3: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Period effects; p = 0.7494, ANOVA
Statistical Analysis 4: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Mixed effects modelling; p = 0.001, Mixed Models Analysis; Mean Difference (Net) = -13.31, 95% CI 2-sided [-21.29 to -5.33]

2. Secondary Outcome: Experience of Pain
Description: A 100mm modified Visual Analogue Scale (VA scale) measuring pain during intraoral scanning taking versus alginate impressions taken in the orthodontic setting. A higher score would indicate a more negative experience. Minimum value: 0, Maximum value: 100
Time Frame: Immediately following intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan | Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions
Number analyzed (Participants) | 42 | 42
score on a scale | -3.5 [-10.75 to 3.71] | -3.3 [-8.31 to 1.76]
Statistical Analysis 1: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — All units of measure reported for this analysis are the mean within-patient differences between alginate and scan VAS scores (i.e. alginate score - scan score); p = 0.1230, Two-period two-treatment crossover ANOVA — From a 2-period 2-treatment crossover ANOVA, taking sequence and period effects into account; Mean Difference (Net) = -3.4, 95% CI 2-sided [-7.71 to 0.91] — This estimation value assumes period and sequence effects are equal between the treatments
Statistical Analysis 2: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Sequence effects; p = 0.8423, ANOVA
Statistical Analysis 3: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Period effects; p = 0.9544, ANOVA

3. Secondary Outcome: Relative Speed of Impression
Description: A 100mm modified Visual Analogue Scale (VA scale) measuring relative speed during intraoral scanning taking versus alginate impressions taken in the orthodontic setting. A higher score would indicate a more negative experience. Minimum value: 0, Maximum value: 100
Time Frame: Immediately following intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan | Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions
Number analyzed (Participants) | 42 | 42
score on a scale | -3.5 [-8.01 to 1.11] | -3.4 [-8.29 to 1.58]
Statistical Analysis 1: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0439, Two-period two-treatment crossover ANOVA — From a 2-period 2-treatment crossover ANOVA, taking sequence and period effects into account; Mean Difference (Net) = -3.4, 95% CI 2-sided [-6.69 to -0.12] — This estimation value assumes period and sequence effects are equal between the treatments
Statistical Analysis 2: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Sequence effects; p = 0.3878, ANOVA
Statistical Analysis 3: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Period effects; p = 0.9772, ANOVA

4. Secondary Outcome: Nausea and/or Coughing
Description: A 100mm modified Visual Analogue Scale (VA scale) measuring nausea and/or coughing during intraoral scanning taking versus alginate impressions taken in the orthodontic setting. A higher score would indicate a more negative experience. Minimum value: 0, Maximum value: 100
Time Frame: Immediately following intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan | Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions
Number analyzed (Participants) | 42 | 42
score on a scale | 12.6 [1.51 to 23.73] | 6.7 [-5.66 to 18.99]
Statistical Analysis 1: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0213, Two-period two-treatment crossover ANOVA — From a 2-period 2-treatment crossover ANOVA, taking sequence and period effects into account; Mean Difference (Net) = 9.6, 95% CI 2-sided [1.50 to 17.79] — This estimation value assumes period and sequence effects are equal between the treatments
Statistical Analysis 2: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Sequence effects; p = 0.1583, ANOVA
Statistical Analysis 3: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Period effects; p = 0.4709, ANOVA

5. Secondary Outcome: Likely Recommendation
Description: A 100mm modified Visual Analogue Scale (VA scale) measuring likely recommendation and/or coughing during intraoral scanning taking versus alginate impressions taken in the orthodontic setting. A higher score would indicate a more negative experience. Minimum value: 0, Maximum value: 100
Time Frame: Immediately following intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan | Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions
Number analyzed (Participants) | 42 | 42
score on a scale | 6.4 [0.22 to 12.66] | 4.1 [-1.74 to 9.96]
Statistical Analysis 1: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0146, Two-period two-treatment crossover ANOVA — From a 2-period 2-treatment crossover ANOVA, taking sequence and period effects into account; Mean Difference (Net) = 5.3, 95% CI 2-sided [1.09 to 9.46] — This estimation value assumes period and sequence effects are equal between the treatments
Statistical Analysis 2: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Sequence effects; p = 0.5911, ANOVA
Statistical Analysis 3: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Period effects; p = 0.5825, ANOVA

6. Secondary Outcome: Ease of Impression for the Operator
Description: A 100mm Visual Analogue Scale (VA scale) measuring ease of impression for the operator during intraoral scanning taking versus alginate impressions taken in the orthodontic setting. A higher score would indicate a more negative experience. Minimum value: 0, Maximum value: 100
Time Frame: Immediately following intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan | Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions
Number analyzed (Participants) | 42 | 42
score on a scale | -1.6 [-11.80 to 8.56] | -8.8 [-15.06 to -2.56]
Statistical Analysis 1: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0817, Two-period two-treatment crossover ANOVA — From a 2-period 2-treatment crossover ANOVA, taking sequence and period effects into account; Mean Difference (Net) = -5.2, 95% CI 2-sided [-11.12 to 0.69] — This estimation value assumes period and sequence effects are equal between the treatments
Statistical Analysis 2: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Sequence effects; p = 0.0910, ANOVA
Statistical Analysis 3: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Period effects; p = 0.2278, ANOVA

7. Secondary Outcome: Confidence Taking the Impression for the Operator
Description: A 100mm Visual Analogue Scale (VA scale) measuring operator confidence during intraoral scanning taking versus alginate impressions taken in the orthodontic setting. A higher score would indicate a more negative experience. Minimum value: 0, Maximum value: 100
Time Frame: Immediately following intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan | Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions
Number analyzed (Participants) | 42 | 42
score on a scale | -1.9 [-6.20 to 2.39] | -2.6 [-6.73 to 1.59]
Statistical Analysis 1: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.1347, Two-period two-treatment crossover ANOVA; From a 2-period 2-treatment crossover ANOVA, taking sequence and period effects into account; Mean Difference (Net) = -2.2, 95% CI 2-sided [-5.17 to 0.69] — This estimation value assumes period and sequence effects are equal between the treatments
Statistical Analysis 2: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Sequence effects; p = 0.9259, ANOVA
Statistical Analysis 3: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Period effects; p = 0.8225, ANOVA

8. Secondary Outcome: Relative Speed of Impression for the Operator
Description: A 100mm Visual Analogue Scale (VA scale) measuring relative speed of impression for the operator during intraoral scanning taking versus alginate impressions taken in the orthodontic setting. A higher score would indicate a more negative experience. Minimum value: 0, Maximum value: 100
Time Frame: Immediately following intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan | Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions
Number analyzed (Participants) | 42 | 42
score on a scale | -8.1 [-21.93 to 5.72] | -14.2 [-27.20 to -1.8]
Statistical Analysis 1: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0200, Two-period two-treatment crossover ANOVA — From a 2-period 2-treatment crossover ANOVA, taking sequence and period effects into account; Median Difference (Net) = -11.2, 95% CI 2-sided [-20.47 to -1.83] — This estimation value assumes period and sequence effects are equal between the treatments
Statistical Analysis 2: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Sequence effects; p = 0.9104, ANOVA
Statistical Analysis 3: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Period effects; p = 0.5194, ANOVA

9. Secondary Outcome: Operator Experience of Sickness or Coughing
Description: A 100mm Visual Analogue Scale (VA scale) measuring operator experience of sickness or coughing during intraoral scanning taking versus alginate impressions taken in the orthodontic setting. A higher score would indicate a more positive experience. Minimum value: 0, Maximum value: 100
Time Frame: Immediately following intervention
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan | Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions
Number analyzed (Participants) | 42 | 42
score on a scale | -26.9 [-38.50 to -15.24] | -19.6 [-29.38 to -9.81]
Statistical Analysis 1: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.00005, Two-period two-treatment crossover ANOVA — From a 2-period 2-treatment crossover ANOVA, taking sequence and period effects into account; Mean Difference (Net) = -23.2, 95% CI 2-sided [-30.71 to -15.75] — This estimation value assumes period and sequence effects are equal between the treatments
Statistical Analysis 2: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Sequence effects; p = 0.1369, ANOVA
Statistical Analysis 3: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Period effects; p = 0.3366, ANOVA

10. Secondary Outcome: Chairside Time Taken to Complete Impression Method
Description: A quantitative time measure will be recorded for each impression method
Time Frame: Immediately following intervention
Measure: Mean (95% Confidence Interval); unit: seconds (within-patient)
Arm/Group | Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan | Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions
Number analyzed (Participants) | 42 | 42
seconds (within-patient) | -88.8 [-136.62 to -41.04] | -151.1 [-185.38 to -116.81]
Statistical Analysis 1: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.00005, Two-period two-treatment crossover ANOVA; From a 2-period 2-treatment crossover ANOVA, taking sequence and period effects into account; Mean Difference (Net) = -120.0, 95% CI 2-sided [-149.54 to -90.38] — This estimation value assumes period and sequence effects are equal between the treatments
Statistical Analysis 2: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Sequence effects; p = 0.8509, ANOVA
Statistical Analysis 3: Comparison: Arm 1 - Alginate Impressions Followed by Digital Intraoral Scan vs Arm 2 - Digital Intraoral Scan Followed by Alginate Impressions; Test type: Superiority — Period effects; p = 0.0355, ANOVA

11. Secondary Outcome: Operator Preference
Description: A simple question to determine operator preference for intraoral scanning versus alginate impressions.
Time Frame: Immediately following completion of participant data collection
Population: This involved asking the 4 operators (clinicians) their overall preference for alginate impressions or intraoral scans during the clinical trial.
Measure: Count of Participants; unit: Participants
Groups:
- Alginate: Preference for alginate
- Intraoral Scan: Preference for intraoral scan
Arm/Group | Alginate | Intraoral Scan
Number analyzed (Participants) | 4 | 4
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events across the 2 days in which they underwent intervention (either intraoral scan or alginate impression). There was a washout period of at least 4 weeks between these 2 days.
Description: Adverse Event (AE) - Any untoward medical occurrence in a participant, including occurrences which are not necessarily caused by or related to study procedures.
  Serious Adverse Event (SAE) - A serious adverse event is any untoward medical occurrence that:
  * results in death
  * is life-threatening
  * requires inpatient hospitalisation or prolongation of existing hospitalisation
  * results in persistent or significant disability/incapacity
  * consists of a congenital anomaly or birth defect
Groups:
- Alginate Impression: Alginate impressions: Alginate impressions are the conventional method of creating dental moulds for orthodontic records. A plastic tray is filled with an alginate material, which is placed into the mouth to take a mould of the teeth. This requires two moulds for both top and bottom arches. In addition, the participant would also bite into a warm piece of wax to record their bite.
Arm/Group | Alginate Impression | Intraoral Scan
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/86
Other Adverse Events (participants affected / at risk) | 0/84 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT05194956/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT05194956/SAP_001.pdf